CLINICAL TRIAL: NCT01460589
Title: Early Commencement of Adjuvant Chemotherapy for Stage III Colon Cancer: a Multicenter Randomized Trial
Brief Title: Early Commencement of Adjuvant Chemotherapy for Colon Cancer
Acronym: ECTX
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Gyu-Seog Choi, Professor, Kyungpook National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KNUHCRC004
Record Dates: First submitted 2011-10-25; First posted 2011-10-27 (Estimated); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colon Cancer
Keywords: colon cancer; Chemotherapy; adjuvant
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- early commencement (Experimental): Individuals who initiate the adjuvant chemotherapy from 10 to 14 days after surgery
  Interventions: Drug: timing to initiate the adjuvant FOLFOX chemotherapy
- conventional commencement (Active Comparator): Individuals who initiate the adjuvant chemotherapy after 14 days after surgery
  Interventions: Drug: timing to initiate the adjuvant FOLFOX chemotherapy

INTERVENTIONS:
Drug: timing to initiate the adjuvant FOLFOX chemotherapy — Chemotherapy regimen: FOLFOX-6, every 2weeks, total 12 cycles treatment day1: Oxaliplatin 85mg/m2 day1: Leucovorin 200mg/m2 day1: 5-FU 400mg/m2 IV bolus and 2,400mg/m2 over 46 hours
  Other Names: early commencement of chemotherapy

SUMMARY:
This study sets up the final study end point and three detailed goals as the following.

The main objective of study: This trial is done to assess the safety and benefit of early adjuvant chemotherapy from 10 to 14 days after surgery compared with conventional commencement after 2weeks for treatment of patients with colon cancer.

Detailed goal of study:

The primary endpoint: This study is designed to assess whether early commencement of adjuvant chemotherapy improves the 3-year disease-free survival, overall survival and recurrence rate.

The secondary endpoint: This study aims to compare short-term cumulative complications between early and conventional commencement of adjuvant chemotherapy after laparoscopic resection of colon cancer. This study will also assess the quality of life and side effects of chemotherapy.

DETAILED DESCRIPTION:
Chemotherapy regimen: FOLFOX-6, every 2weeks, total 12 cycles treatment

* day1: Oxaliplatin 85mg/m2
* day1: Leucovorin 200mg/m2
* day1: 5-FU 400mg/m2 IV bolus

  * 2,400mg/m2 over 46 hours

ELIGIBILITY:
Inclusion Criteria:

* Eligibility rule of enrollment
* Rectal adenocarcinoma that were 15 cm or more from the anal verge
* pathologically diagnosed stage II or III disease
* patients who meet the discharge criteria within 10days after surgery
* Patients with adequate hepatic, renal, and bone marrow function, and a left ventricular ejection fraction of 55% or higher measured by echocardiography

Exclusion Criteria:

* An ineligibility to participate in the clinical study based on the judgment of investigators from a legal perspective
* A past history of chemotherapy
* tumor with obstruction or perforation
* tumor with distant metastases
* synchronous tumor
* relative or absolute contraindications of chemotherapy
* Recent MI, CVA, nitrate medication
* Severe cardiovascular disease, psychiatric disease
* Severe hepatic dysfunction (GOT, GPT ≥100IU/L)
* Renal dysfunction (Cr ≥2mg/dl)
* The concurrent presence of other severe medical diseases

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2013-01-13 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
3-year disease free survival rate | up to 3 years after operation
  A survival analysis will be performed using the Kaplan-Meier method, for which a comparison of the survival curve will also made using a Log-rank test.

SECONDARY OUTCOMES:
short-term cumulative surgery-related complications during chemotherapy | up to 26 weeks after operation
  A comparison of the postoperative recovery variables, the postoperative complications and mortality
side effects of chemotherapy | during chemotherapy period
  check Anemia, Leukopenia, Neutropenia, Thrombocytopenia, Edema, Fever, Insomnia, Asthenia, Anorexia, Nausea, Vomiting, Constipation, Diarrhea, Hand foot syndrome, Dyspepsia, Creatinine, AST, ALT, Bilirubin, abdominal pain, GI bleeding, diarrhea

CONTACTS AND LOCATIONS:
Overall Officials: Jun Seok Park, M.D.Ph.D, Study Chair — Kyunpook National Univercity Medical Center
Locations (2):
- South Korea (2):
  - Kyungpook National University Medical center, Daegu
  - Jun Seok Park, Daegu